CLINICAL TRIAL: NCT06900296
Title: ImmuNe ParameTERs to Predict Immunotherapy REsponse and Toxicity (INTERPRET)
Acronym: INTERPRET
Status: Not yet recruiting | Type: Observational
Sponsor: Indiana University (Other)
Collaborators: Indiana Institute of Personalized Medicine (Unknown)
Responsible Party: Principal Investigator, Tyler Andrew Shugg, Assistant Professor, Indiana University
Other Study IDs: PHARM-IUSCCC-0913
Record Dates: First submitted 2025-03-21; First posted 2025-03-28 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Cancer
Keywords: immunotherapy treatment
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — This study is observational in nature and will involve no medical interventions outside of collecting 1-10 blood samples at 1-10 separate study visits
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a prospective observational study that will collect blood samples at 1-10 timepoints related to initiation of immunotherapy. The study may collect samples before the start of immunotherapy and/or at clinically significant timepoints during immunotherapy treatment.

DETAILED DESCRIPTION:
The long-term goal of this research is to identify immunologic and other blood-borne markers of immunotherapy efficacy and toxicity. The objective of this proposal is to identify associations between immunologic parameters and other blood-borne markers with treatment response, irAE development, or relevant biomarkers of both outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years old at the time of informed consent.
2. Have a diagnosis of cancer and initiating therapy with single agent or combination therapy that includes an immunotherapy (see Appendix 16.1 for list of immunotherapy classes).
3. Ability to provide written informed consent and HIPAA authorization.

Exclusion Criteria:

1. Not meeting any of the previously described inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults diagnosed with cancer and initiating immunotherapy treatment
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2026-05 (Estimated); Primary Completion 2029-04 (Estimated); Study Completion 2029-04 (Estimated)

PRIMARY OUTCOMES:
Quantification of plasma concentrations | through study completion (i.e. up to 12 months)
  Including cytokines, chemokines, growth factors, and other relevant immunologic molecules from blood samples
Profiling of immune cells | through study completion (i.e. up to 12 months)
  Plasma concentrations of immunologic molecules will be assayed using immunoassays or plasma proteomic approaches. Profiling of immune cells will be performed using flow cytometry, RNA sequencing, and other established approaches.

SECONDARY OUTCOMES:
Assessment of genomic variants | through study completion (i.e. up to 12 months)
  Whole genome sequencing of germline DNA isolated from blood samples.

CONTACTS AND LOCATIONS:
Overall Officials: Tyler Shugg, PharmD, PhD, Principal Investigator — Indiana University
Locations (1):
- Indiana University Melvin and Bren Simon Comprehensive Cancer Center, Indianapolis, Indiana, United States